CLINICAL TRIAL: NCT02290197
Title: Knee Dislocation - Clinical Evaluation of the Use of Hinged External Fixator After Ligament Reconstruction. Randomized Prospective Study.
Brief Title: Knee Dislocation - Clinical Evaluation of the Use of Hinged External Fixator After Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Fábio Janson Angelini, Assistant Physician, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0886-09
Record Dates: First submitted 2014-10-29; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Knee Dislocation
MeSH Terms: conditions — Knee Dislocation | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hinged External Fixator (Experimental): Hinged external fixator allows early and aggressive joint mobility in the sagittal plane only. Flexion and extension are permitted, but rotational movements, translations in the anterior-posterior plane, lateral (varus) and medial (valgus) openings are not allowed. Thus protective stability is ensured for ligament reconstruction procedures. Simultaneously we allow immediate joint mobilization, reducing the risk of arthrofibrosis, joint stiffness and postoperative ligament laxity.
  Interventions: Procedure: Surgery; Device: Hinged External Fixator
- Cast Immobilization (Active Comparator): In these patients we used cast postoperatively for 3 weeks. After this period we use a removable bracing and initiate rehabilitation with physical therapy.
  Interventions: Procedure: Surgery; Device: Cast Immobilization

INTERVENTIONS:
Procedure: Surgery — Surgical reconstruction of all injured ligaments.
Device: Hinged External Fixator — Hinged external fixator is used postoperatively for 6 weeks. Early joint mobility in the sagittal plane is encouraged.
  Arms: Hinged External Fixator
Device: Cast Immobilization — Cast is used postoperatively for 3 weeks. After this period we use a removable bracing and initiate rehabilitation with physical therapy.
  Arms: Cast Immobilization

SUMMARY:
Knee dislocation is a serious injury, usually caused by high-energy trauma. It is classically defined as complete loss of articular congruence between the femur and the tibia, confirmed by radiography. However it is common that the reduction happens spontaneously. For this reason, today the investigators also consider a patient suffered knee dislocation in the presence of multi-ligament injury involving the posterior cruciate ligament, often in association with anterior cruciate ligament, lateral and/or medial ligamentous complex.

It is considered a serious injury, because both the strong association with vascular and nerve damage, which can lead to the need for limb amputation, such as the difficulty in obtaining a good functional outcome even after treatment of all ligament injuries.

The treatment of these injuries aims to achieve knee stability. Joint mobility is often sacrificed in the postoperative period, with the use of immobilizations such as casts, splints or bracing. Unfavorable clinical outcomes with high rates of stiffness and joint pain are very common in these patients. In attempts to improve these results, rehabilitation protocols with early range of motion can be employed. However, results may remain unsatisfactory, predominantly because of knee instability recurrence.

Stannard and Zaffagnini proposed a new model for treatment of acute knee dislocations. In this model, after multi-ligament reconstruction or repair, a knee articulated external fixator is used. Such external fixator allows early and aggressive joint mobility in the sagittal plane only. Flexion and extension are permitted, but rotational movements, translations in the anterior-posterior plane, lateral (varus) and medial (valgus) openings are not allowed. Thus protective stability is ensured for ligament reconstruction procedures. Simultaneously the investigators allow immediate joint mobilization, reducing the risk of arthrofibrosis, joint stiffness and postoperative ligament laxity.

There is no consensus regarding the use of hinged external fixator postoperatively in multiple ligament reconstruction procedures for treatment of knee dislocations.

The objective of this study is comparing functional outcomes after ligament reconstruction in patients with knee dislocation, with or without the use of hinged external fixator.

ELIGIBILITY:
Inclusion Criteria:

* adults aged between 18 and 50 years old, diagnosed with knee dislocation, classified as KD-III and KD-IV
* absence of knee arthritis in initial radiographs
* absence of systemic diseases or disorders of collagen altering bone quality
* absence of previous surgical interventions in the knee
* possibility of using medications
* maximum of three months of injury to treatment
* understanding and acceptance by the patient to participate

Exclusion Criteria:

* abandoning medical care
* inability to follow the treatment plan

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Knee stability | 12 months postoperative
  Physical examination performed by an independent investigator (Physical Therapist).
  Evaluation of posterior drawer according to the IKDC objective criteria: A (normal - 0 to 2mm); B (near normal - 3 to 5 mm); C (abnormal - 6 to 10mm); D (severely abnormal - greater than 10mm).
  Evaluation of the posterior lateral corner according to the IKDC objective - External Rotation Test (patient in prone position, knee flexed 90 degrees). A (normal - < 5 degrees); B (near normal - 6 to 10 degrees); C (abnormal - 11 to 19 degrees); D (severely abnormal - greater than 20 degrees)

SECONDARY OUTCOMES:
Range of motion | 12 months postoperative
  Physical examination performed by an independent investigator (Physical Therapist).
  Knee range of motion (flexion / extension) in degrees.
Pain | 12 months postoperative
  Visual Analogue Scale - VAS
IKDC | 12 months postoperative
  Clinical score
Lysholm | 12 months postoperative
  Clinical score
Adverse events | 12 months postoperative
  Adverse events from surgery or rehabilitation period

CONTACTS AND LOCATIONS:
Overall Officials: Fabio J Angelini, M.D., Principal Investigator — University of Sao Paulo; Roberto F Mota e Albuquerque, Ph.D., Study Director — University of Sao Paulo; Gilberto L Camanho, Ph.D., Study Chair — University of Sao Paulo
Locations (1):
- Hospital das Clinicas - University of Sao Paulo, São Paulo, São Paulo, Brazil